CLINICAL TRIAL: NCT03072953
Title: A Phase 2a, Open-label, Proof of Concept Study to Determine the Efficacy and Safety of Etrasimod (APD334) in Patients With Pyoderma Gangrenosum
Brief Title: Efficacy and Safety of APD334 in Patients With Pyoderma Gangrenosum
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated [Sponsor decision to terminate the study]
Sponsor: Arena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APD334-011
Record Dates: First submitted 2017-02-17; First posted 2017-03-08 (Actual); Results first posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — etrasimod

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- APD334 (Other): APD334 active treatment for 12 weeks.
  Interventions: Drug: APD334

INTERVENTIONS:
Drug: APD334 — APD334 active treatment
  Other Names: Etrasimod

SUMMARY:
The purpose of this Phase 2a, open label, proof-of-concept clinical study is to assess the efficacy and safety of etrasimod (APD334) in patients with Pyoderma Gangrenosum.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female (18-80 years).
2. Able to provide a signed informed consent prior to any study related procedure being conducted.
3. Diagnosis of PG with active, non-healing ulcer.
4. Considered to be in stable health in the opinion of the investigator as determined by:

   1. A screening physical examination with no clinically significant abnormalities unrelated to PG.
   2. Vital signs at screening: pulse rate ≥ 55 bpm, systolic blood pressure ≥ 90 mmHg, and diastolic blood pressure ≥ 55 mmHg.
   3. Liver function tests (alanine aminotransferase/aspartate aminotransferase, bilirubin and alkaline phosphatase) < 2x the upper limit of normal.
   4. All other pre-study clinical laboratory findings within normal range, or if outside of the normal range are not deemed clinically significant in the opinion of the investigator with exemption to leucopenia and lymphopenia - please refer to exclusion criterion 24.
   5. No clinical abnormalities noted in the12-lead electrocardiogram in the opinion of the investigator (Refer also to exclusion criterion 13).
   6. No evidence of macular edema in an ophthalmology evaluation (performed by an ophthalmologist), supported with optical coherence tomography, where available (dependent on site capability) at screening.
5. Eligible male and female participants must agree not to participate in a conception process (i.e. active attempt to let female partner to become pregnant or to impregnate, sperm donation, oocyte donation, in vitro fertilization) for at least 30 days after the last dose of study drug.

Non-sterile participants who are sexually active must take adequate contraception measures.

Exclusion Criteria:

1. Clinically significant infection as judged by the investigator with an end date less than 6-weeks prior to treatment start (Day 1). In case of infection requiring hospitalization or intravenous antimicrobial therapy, or opportunistic infection, this infection must have ended at least 8 weeks prior to Day 1.
2. Infection with hepatitis C virus anytime in the past; confirmed active infection with hepatitis B virus at screening.
3. History of severe renal or severe hepatic impairment.
4. Current active or latent tuberculosis (TB).
5. A positive diagnostic TB test at screening.
6. Exposure to B-cell or T-cell targeted therapies (such as natalizumab, rituximab, abatacept) within 5 half-lives prior to Day 1.
7. Exposure to other immunosuppressive, immunomodulating or antineoplastic agents.
8. Receipt of any investigational agent within 30 days or 5 half lives (whichever is longer), prior to Day 1.
9. Use of moderate to strong inhibitors of CYP2C9.
10. Abnormal forced expiratory volume (FEV1) or forced vital capacity (FVC).
11. Any known history of congenital or acquired immuno-deficiency.
12. Recent history (within 6 months of screening visit) of cardio- or cerebrovascular disease, acute coronary syndrome, myocardial infarction, unstable angina, cerebro-vascular accident, including transient ischemic attack.
13. History or presence of cardiac arrhythmia, conduction system disease, or use of Class Ia or Class III anti arrhythmic agents, or baseline QTc ≥ 500 msec.
14. Congestive heart failure (NYHA III or NYHA IV)
15. Any surgical procedure requiring general anesthesia within 30 days prior to Day 1 or plans to undergo major surgery during the study period.
16. History of retinal macular edema.
17. History of or signs and symptoms of progressive multifocal leukoencephalopathy (PML) as assessed by the PML checklist at screening.
18. History of more than one episode of herpes zoster or any episode of disseminated zoster.
19. Participants without documented positive varicella zoster virus (VZV) IgG antibody status or participants who have not completed VZV vaccination within 6 weeks prior to Day 1.
20. Receipt of live vaccine within 6 weeks prior to Day 1.
21. History of lymphoproliferative disorder, lymphoma, leukemia, myeloproliferative disorder, or multiple myeloma.
22. History of malignancy except for adequately treated basal cell skin cancer and in situ carcinoma of the cervix of the uterus that have been completely excised with documented, clear margins.
23. History of severe allergic or anaphylactic reactions requiring medical attention.
24. Leukopenia or lymphopenia at screening.
25. Current or recent history (within 1 year prior to Day 1) of alcohol dependence or illicit drug use.
26. Active psychiatric problems that, in the investigator's opinion, may interfere with compliance with the study procedures.
27. History of any other clinically significant medical condition that, in the investigator's opinion, would preclude participant from safe participation in the study.
28. Inability to attend all the study visits or comply with study procedures.
29. Prior exposure to etrasimod (APD334) or prior participation in any study of etrasimod (APD334).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arena CT.gov Administrator, Study Director — Arena Pharmaceuticals
Locations (6):
- Australia (5):
  - Westmead Hospital, Westmead, New South Wales
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Eastern Clinical Research Unit, Box Hill, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
- Braemar Day Hospital, Hamilton, New Zealand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- APD334: During the 12-week treatment period, participants received etrasimod active treatment, administered orally, once daily.
Period: Overall Study
Arm/Group | APD334
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | APD334
Number analyzed (Participants) | 2
Age, Customized [Count of Participants; unit: Participants]
  Between 18 to 80 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Reporting demographic results for this study in which only two participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported.
  Male | NA — Reporting demographic results for this study in which only two participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | NA — Reporting demographic results for this study in which only two participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported.
  Not Hispanic or Latino | NA — Reporting demographic results for this study in which only two participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported.
  Unknown or Not Reported | NA — Reporting demographic results for this study in which only two participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Exploratory Endpoint - Change From Baseline in Physician Global Assessments for Active Skin Manifestations
Description: The physician's global assessment for active skin manifestations recorded the number of ulcers, target lesion noted for endpoint evaluation, diameters of each target lesion and score of evaluation at each visit. The scores ranged from 0 (total resolution) to 4 (no evidence of healing).
Time Frame: Week 12
Population: Efficacy analyses were not conducted due to low enrollment (N=2). In order to protect participant's privacy, the results from the enrolled participants cannot be reported.
Arm/Group | APD334
Number analyzed (Participants) | 0

2. Primary Outcome: Exploratory Endpoint - Change From Baseline in Patient Global Assessments for Active Skin Manifestations
Description: The patient global assessment for active skin manifestation recorded the disease and pain severity using a visual analogue to mark the participant's score. Participants were asked to rate their disease severity from "not severe" to "extremely severe" and pain levels from "no pain at all' to "worst pain imaginable" in the past one week.
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | APD334
Number analyzed (Participants) | 0

3. Primary Outcome: Exploratory Endpoint - Change From Baseline in Dermatology Life Quality Index (DLQI) Score
Description: The DLQI questionnaire assessed how much a participant's life is affected through their skin problem in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure and sport activities, work or school activities, personal relationships and treatment- related feelings. Participants responded to the 10 questions on a scale from 0 (not at all) to 3 (very much) with a total score ranging from 0 to 30. Higher scores indicated that the skin problem had an extremely large effect on the participant's life whereas lower scores indicated that the disease has minimal to no effect at all.
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | APD334
Number analyzed (Participants) | 0

4. Primary Outcome: Exploratory Endpoint - Change From Baseline in C-reactive Protein Levels
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | APD334
Number analyzed (Participants) | 0

5. Primary Outcome: Exploratory Endpoint - Assessments of Target Lesions
Description: Changes in surface area
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | APD334
Number analyzed (Participants) | 0

6. Primary Outcome: Exploratory Endpoint - Assessment of Punch Biopsies
Description: Changes in histology.
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | APD334
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Number of Participants With Adverse Events and Clinically Significant (CS) Safety Measurements
Description: Safety was assessed by monitoring and recording all adverse events, clinical laboratory tests (including hematology, serum chemistry, coagulation, and urinalysis), physical and neurological examinations, vital sign measurements, and 12-lead electrocardiograms. The number of participants with adverse events and CS safety measures have been reported.
Time Frame: Up to approximately 12 weeks
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | APD334
Number analyzed (Participants) | 2
Participants
  Adverse events | 2
  CS clinical laboratory values | 0
  CS physical & neurological examinations | 0
  CS vital sign measurements | 0
  CS 12-lead ECG measurements | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 12 weeks
Arm/Group | APD334
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | APD334 (N=2)
Diarrhea (Gastrointestinal disorders) | 1
headache (Nervous system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Sore hip (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
Due to limited enrollment (N=2), this clinical trial was terminated by the Sponsor and no efficacy analyses were conducted. To protect the participant's privacy, demography and efficacy data are not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/53/NCT03072953/Prot_SAP_000.pdf